CLINICAL TRIAL: NCT02389751
Title: GUARDIAN-1 Trial: A Phase 1 Study of Ganetespib in Combination With Chemoradiation for Stage II-III Esophageal Carcinoma
Brief Title: Ganetespib in Combination With Paclitaxel, Carboplatin, and Radiation Therapy in Treating Patients With Stage II-III Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0815; NCI-2015-00492 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0815 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Malignant Neoplasm of the Cervical Esophagus; Malignant Neoplasm of the Thoracic Esophagus; Stage IIA Esophageal Cancer AJCC v7; Stage IIB Esophageal Cancer AJCC v7; Stage IIIA Esophageal Cancer AJCC v7; Stage IIIB Esophageal Cancer AJCC v7; Stage IIIC Esophageal Cancer AJCC v7
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Carboplatin; STA 9090; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ganetespib, paclitaxel, carboplatin, radiation) (Experimental): Patients receive ganetespib IV over 1 hour, paclitaxel IV over 1 hour, and carboplatin IV over 30 minutes once a week on day 1. Patients also undergo radiation therapy 5 days a week for 5.5 weeks or for a total of 28 treatments. Treatment continues for 28 treatment days (5.5 weeks) in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Carboplatin; Drug: Ganetespib; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Ganetespib — Given IV
  Other Names: Hsp90 Inhibitor STA-9090; STA-9090
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of ganetespib when given together with paclitaxel, carboplatin, and radiation therapy in treating patients with stage II-III esophageal cancer. Ganetespib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving ganetespib in combination with paclitaxel, carboplatin, and radiation therapy may be a better treatment for patients with esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated disease (MTD) and the recommended phase II dose of ganetespib to combine with standard carboplatin and paclitaxel chemotherapy and radiotherapy in stage II-III patients with esophageal carcinoma.

SECONDARY OBJECTIVES:

I. To assess the response rate based on fludeoxyglucose-positron emission tomography/computed tomography (FDG-PET/CT) +/- CT with contrast imaging response assessment after completion of chemoradiation.

II. To determine the 1 year overall survival (OS) rate. III. To determine the progression-free survival (PFS) rate. IV. To determine the pathologic complete response (pCR) rate for patients who undergo surgery.

OUTLINE: This is a dose-escalation study of ganetespib.

Patients receive ganetespib intravenously (IV) over 1 hour, paclitaxel IV over 1 hour, and carboplatin IV over 30 minutes once a week on day 1. Patients also undergo radiation therapy 5 days a week for 5.5 weeks or for a total of 28 treatments. Treatment continues for 28 treatment days (5.5 weeks) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma or squamous cell carcinoma of the cervical esophagus, thoracic esophagus, or gastroesophageal junction
* Stage II or III esophageal carcinoma according to the American Joint Committee on Cancer (AJCC) 7th edition staging
* Esophagogastroduodenoscopy (EGD) with endoscopic ultrasound (EUS) +/- biopsy at M.D. Anderson are required to confirm staging
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Patients should have no contraindications for chemotherapy or radiation, and should receive either definitive chemoradiation therapy or preoperative chemoradiation therapy
* Patients must have received baseline FDG-PET/CT +/- CT with contrast within 1 month +/- 2 weeks prior to study entry, and should have no contraindications to PET or CT imaging
* Women of child-bearing potential and men must agree to adequate contraception (hormonal or barrier method of birth control; abstinence) during and up to 30 days after discontinuing treatment
* Women of child-bearing potential must have a negative serum pregnancy test within 14 days of study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* White blood cells (WBC) >= 2500 cells/ul
* Hemoglobin >= 9 g/dL
* Platelets >= 100x10^9/L
* Albumin >= 2.5 g/dL
* Serum bilirubin =< 1.5x institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 x institutional ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x institutional ULN
* Baseline screening corrected QT (QTc) < 470 ms is eligible

Exclusion Criteria:

* Prior radiation to the chest or abdomen
* Previous or concomitant malignancy - EXCEPTIONS: patients with curatively treated carcinoma in situ of the cervix, basal cell of the skin, transitional cell carcinoma of the bladder, or early stage cancers at non-overlapping sites with no evidence of disease for >= 3 years
* No induction chemotherapy
* Pregnant or breast-feeding females; patients who become pregnant during active therapy will be immediately removed from the study
* Uncontrolled intercurrent illness or serious medical conditions including, but not limited to:

  * Clinically significant, uncontrolled, major cardiac, respiratory, renal, hepatic, gastrointestinal, or hematologic disease
  * Active uncontrolled infection
  * Symptomatic congestive heart failure, unstable angina, or cardiac dysrhythmia not controlled by pacer device
  * No myocardial infarction within 3 months of registration
  * Symptomatic inflammatory bowel disease with uncontrolled diarrhea
* Major cardiac-related diseases, medications, or laboratory abnormalities including the following: a) clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling temporary pacemaker, b) ventricular tachycardia or a supraventricular tachycardia that requires treatment with a class Ia antiarrhythmic drug (eg, quinidine, procainamide, disopyramide) or class III antiarrhythmic drug (eg, sotalol, amiodarone, dofetilide); use of other antiarrhythmic drugs is permitted; c) use of medications that have been linked to the occurrence of torsades de pointes, d) second- or third-degree atrioventricular (AV) block unless treated with a permanent pacemaker, e) complete left bundle branch block (LBBB), f) history of long QT Syndrome or a family member with this condition, g) if baseline QTc > 470 ms, average of triplicate electrocardiogram (ECG) recordings is necessary; if average value of QTc is > 470 ms, patient is ineligible for the study; h) serum potassium, magnesium, and calcium levels outside the laboratory's reference range
* Known immediate or delayed hypersensitivity reaction to carboplatin, paclitaxel, polysorbate 80, or any other component of the formulation
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to study registration, and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to registration
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) either preceding the first dose of ganetespib or during the study period
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited: a) other anti-cancer therapy while on study treatment, b) the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* Known human immunodeficiency virus (HIV), active hepatitis B virus (HBV), or active hepatitis C virus (HCV) infection (with the exception of chronic or cleared HBC and HCV infection, which will be allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
MTD and recommended phase II dose of ganetespib, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 70 days
  The MTD is defined as the dose for which the posterior mean probability of dose-limiting toxicity is closest to 30%.

SECONDARY OUTCOMES:
Response rate based on FDG-PET/CT +/- CT imaging response assessment after completion of chemoradiation | At 6 weeks after completion of chemoradiation therapy
OS | Up to 5 years
PFS | Up to 5 years
pCR for patients who undergo surgical resection after neoadjuvant therapy | Up to 10 weeks after completion of chemoradiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org